CLINICAL TRIAL: NCT05916638
Title: Role of Monocytes (Mo) and Macrophages (Ma) in Sarcoidosis and in Tuberculosis
Brief Title: MoMa Signature During Granulomatosis
Acronym: MOSAR
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230273; 2022-A02637-36 (Other: IDRCB)
Record Dates: First submitted 2023-05-17; First posted 2023-06-23 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Sarcoidosis; Tuberculosis
Keywords: tuberculosis; sarcoidosis; granuloma; monocytes; macrophages
MeSH Terms: conditions — Sarcoidosis; Tuberculosis; Granuloma | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, lung biopsy and Bronchoalveolar fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sarcoidosis: patients diagnosed with sarcoidosis
  Interventions: Other: blood sample
- Tuberculosis: patients diagnosed with tuberculosis
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample — blood sample collection

SUMMARY:
Sarcoidosis is a systemic inflammatory disease characterized by unspecific granuloma formation. Our hypothesis is that granuloma formation and maintenance mainly relies on the overactivation of monocytes (Mo) and macrophages (Ma). To this end, the study aims (i) to define MoMa systemic signature in sarcoidosis, (ii) to characterize this signature in situ on tissue samples, and (iii) to identify causative factors that participate to the MoMa chronic overactivation. Thus, a cohort of sarcoidosis patients will be compared with tuberculosis patients. The MoMa systemic signature will be defined on whole blood (TruCulture model) and then in situ through different methods (multi-parameter spectral flow cytometry, RNA-seq, Luminex, imaging mass cytometry). The epigenome of monocytes will be studied thanks to CUT&Tag. The MoMa systemic signature will be defined ex vivo at different time points during the course of the disease with phenotypic, transcriptomic, cytokine and functional approaches. The previously identified signature will be studied in situ and completed by the characterization of granuloma architecture and microenvironmental interactions, which could be modulated by epigenetic modifications. Hence, the epigenome of monocytes will be analyzed in two groups (sarcoidosis and tuberculosis). These results would allow to better understand sarcoidosis physiopathology and, in fine, may raise new therapeutic strategies. Finally, the study could challenge the dogma on innate immunity/auto-inflammation versus adaptive immunity/auto-immunity/memory.

DETAILED DESCRIPTION:
"Sarcoidosis is an inflammatory disease characterized by the presence of coalescing, tightly clustered, non-necrotizing granulomas. The diagnosis is based on three major criteria: a compatible clinical presentation, the presence of non-necrotizing granulomatous inflammation, and the exclusion of alternative granulomatous diseases. A wide range of clinical phenotypes are observed depending on the location of the granulomatous lesions which can affect any organ, with the lungs being the most affected site. Sarcoidosis shares many similarities with tuberculosis, in which granuloma formation is triggered by Mycobacterium tuberculosis (M. tb). These phenotypic similarities between the two diseases present many challenges for diagnosis, clinical management and therapy.

Our understanding of the factors that contribute to sarcoidosis development, granuloma formation and maintenance remains limited. Part of this challenge is that granuloma development may involve both environmental and genetic factors, which contribute to the recruitment of immune cells to form the granuloma. Immune cells involved in the granuloma include (1) CD4 Th1 and Th17 T cells and their associated cytokines (e.g, IFNγ, TNFα, IL-17, IL-2); and (2) monocytes (Mo) and macrophages (Ma) including proinflammatory M1 and pro-fibrosis M2 types. However, the specific factors that contribute to granuloma maintenance and evolution remain to be identified. Among them, we can hypothesized that trained immunity, persistence of the antigen, or the microenvironment are involved in this chronic dysregulated immune response. Such an improved understanding of the pathophysiology of the disease may allow development of new treatments, as currently corticosteroids remain the mainstay of therapy.

Our main hypothesis is that granuloma formation and maintenance mainly relies on the overactivation of monocytes (Mo) and macrophages (Ma). To this end, the study aims (i) to define MoMa systemic signature in sarcoidosis, (ii) to characterize this signature in situ on tissue samples, and (iii) to identify causative factors that participate to the MoMa chronic overactivation. Thus, a cohort of sarcoidosis patients will be compared with tuberculosis patients. The MoMa systemic signature will be defined on whole blood (TruCulture model) and then in situ through different methods (multi-parameter spectral flow cytometry, RNA-seq, Luminex, imaging mass cytometry). The epigenome of monocytes will be studied thanks to CUT&Tag. The MoMa systemic signature will be defined ex vivo at different time points (M0, M6 and M12) during the course of the disease with phenotypic, transcriptomic, cytokine and functional approaches. The previously identified signature will be studied in situ and completed by the characterization of granuloma architecture and microenvironmental interactions, which could be modulated by epigenetic modifications. Hence, the epigenome of monocytes will be analyzed in two groups (sarcoidosis and tuberculosis). These results would allow to better understand sarcoidosis physiopathology and, in fine, may raise new therapeutic strategies. Finally, the study could challenge the dogma on innate immunity/auto-inflammation versus adaptive immunity/auto-immunity/memory."

ELIGIBILITY:
Inclusion criteria:

1. Male and female > 18 years old
2. Diagnosis of sarcoidosis and of tuberculosis
3. Affiliated to medical insurance

Exclusion criteria:

1. HIV infection
2. pregnant or breastfeeding woman
3. Patient under legal protection, guardianship or curators
4. Absence of signed consent"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with sarcoidosis or tuberculosis
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
macrophage activation in sarcoidosis measured by epigenomic | up to 12 months of follow-up.
  performed on peripheral blood mononuclear cells (PBMCs) isolated from peripheral blood
monocyte activation in sarcoidosis measured by epigenomic | up to 12 months of follow-up.
  performed on peripheral blood mononuclear cells (PBMCs) isolated from peripheral blood
macrophage activation in sarcoidosis measured by flow cytometry | up to 12 months of follow-up.
  performed on peripheral blood mononuclear cells (PBMCs) isolated from peripheral blood
monocyte activation in sarcoidosis measured by flow cytometry | up to 12 months of follow-up.
  performed on peripheral blood mononuclear cells (PBMCs) isolated from peripheral blood
monocyte activation in sarcoidosis measured by transcriptomic | up to 12 months of follow-up.
  performed on peripheral blood mononuclear cells (PBMCs) isolated from peripheral blood
macrophage activation in sarcoidosis measured by transcriptomic | up to 12 months of follow-up.
  performed on peripheral blood mononuclear cells (PBMCs) isolated from peripheral blood
macrophage activation in sarcoidosis measured by cytokine measurement | up to 12 months of follow-up.
  performed on peripheral blood mononuclear cells (PBMCs) isolated from peripheral blood
monocyte activation in sarcoidosis measured by cytokine measurement | up to 12 months of follow-up.
  performed on peripheral blood mononuclear cells (PBMCs) isolated from peripheral blood

SECONDARY OUTCOMES:
monocyte activation in tuberculosis measured by epigenomic | up to 12 months of follow-up.
Identification of a pathogen that triggers sarcoidosis development by metagenomic study | Samples collected before treatment/at diagnosis
identification of epigenetic modifications of monocytes by CUT&Tag method | 12 months of follow-up.
  CUT&Tag-sequencing, also known as cleavage under targets and tagmentation, is a method used to analyze protein interactions with DNA
Identification of a diagnostic test to discriminate sarcoidosis and tuberculosis | Samples collected before treatment/at diagnosis
  measurement of IFNγ secretion by whole blood in response to stimulation by tuberculosis antigen

CONTACTS AND LOCATIONS:
Overall Officials: Karim SACRE, MD-PhD, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Bichat, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided